CLINICAL TRIAL: NCT03709459
Title: Impact of the Daily Doxycycline Pre-exposure Prophylaxis (PrEP) on the Incidence of Syphilis, Gonorrhoea and Chlamydia
Acronym: Syphilaxis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kirby Institute (Other Government)
Collaborators: South Australian Health and Medical Research Institute (Other); Monash University (Other)
Responsible Party: Sponsor
Other Study IDs: PHIRG1901
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: STIs Prevention
Keywords: Syphilis, Gonorrhea, Chlamydia, Doxycycline, PrEP, Syphilaxis
MeSH Terms: conditions — Syphilis; Gonorrhea; Chlamydia Infections | interventions — Doxycycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — oropharynx and rectum swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Doxycycline — Participants will be asked to take Doxycycline 100mg/day for 12months duration

SUMMARY:
1. This study is a non-randomized observational cohort trial using before and after comparison to evaluate intervention 2. It would mimic the conditions that would occur outside a clinical trial. 2. After consent and enrolment, all procedures will be guided by the Australian STI Management Guidelines.

3. All enrolling participants will be offered daily doxycycline 100mg 4. All participants will be invited to complete a survey in every 3 months time for 12 months dated from participation.

5. All follow-up information will be collected through electronic data capture to allow accurate and timely analyses.

6. Data collection will be from (i) medical records (ii) online self-completed questionnaire

DETAILED DESCRIPTION:
The last decade has seen increasing rates of bacterial STIs in Australia in gay and bisexual men in particular. Although STIs are easy to diagnose and treatment is effective, untreated STIs can cause significant health issues.

Previous research has shown that taking two100mg doxycycline tablets within 24 hours of sex as prophylaxis reduces syphilis and chlamydia significantly. Also a pilot trial conducted in the US suggested that using 100mg doxycycline as prophylaxis reduced the incidence of gonorrhoea, syphilis and chlamydia. Thus the question of whether taking doxycycline daily in high risk population would reduce the rate of STIs arose.

We set up this study as a non-randomized observational cohort trial using a before and after comparison to evaluate if taking 100mg doxycycline daily would help high risk gay and bisexual men to reduce the possibility of acquiring gonorrhoea, syphilis and chlamydia. Our primary objectives are to:assess acceptability of a daily dosing regimen for doxycycline prophylaxis, and measure the efficacy of 100mg daily doxycycline STI prophylaxis against reinfection with gonorrhoea, chlamydia and syphilis. Our secondary objectives are to: describe patterns of doxycycline use and medication adherence to the recommended schedule participants; evaluate change in behavioral among all study participants; evaluate resistance in the gut microbiota and in those colonized by S aureus at baseline and end of study, in a subset of consenting participants.

The study will be conducted in 3 sexual health centres. Eligible participants will undergo standard care in their trimonthly visit recommended by STI testing guideline, and complete informed consent and a baseline survey. They will be given daily dose of 100mg oral doxycycline for 3 months during the visit, and instruction of how to take the medicine. Questionnaires will be sent out to participants in every 3 months electronically and data will be collected and stored directly into the study survey database. Each participant will be follow-up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or transgender
* Aged 18 years or over
* Reports sex with men in last 3 months
* At least two screenings for syphilis, gonorrhoea and chlamydia in the past 12 months
* A diagnosis of syphilis within the last 12 months, OR a diagnosis of any 2 STIs within the last 12 months and syphilis within the last 24 months.
* HIV +ve, OR HIV -ve and on PrEP for at least 6 months.

Exclusion Criteria:

* Documented or self-reported hypersensitivity to doxycycline or antimicrobial agents from tetracycline family
* A known diagnosis of myasthenia gravis
* Factors or conditions that may compromise a participant's access to health services for follow-up (incarceration or planned relocation that would impact upon proximity to a trial site).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men who report male to male sex in the last 3 months and who have had at least two screening for syphilis, chlamydia and gonorrhoea in the last 12 months, and at least once incidence of syphilis in the last two years, are eligible for the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2024-07-17 (Estimated); Study Completion 2024-12-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of STI (gonorrhoea, chlamydia and infectious syphilis) per 100 person years among study participants | 1 year after the last participant complete their last follow-up visit
  measured using data collected by the ACCESS study
Patterns of daily doxycycline use and adherence to the medication schedule | 1 year after the last participant complete their last follow-up visit
  measured among participants consenting to the adherence and behavioural online survey

SECONDARY OUTCOMES:
Evidence of clinically significant antibiotic resistance in in a subset of participants | 1 year after the last participant who's recruited from the Melbourne site
  including those who do contract STIs during the study and those who don't
Behavioural risk practices among study participants | 1 year after the last participant complete their last follow-up visit
  in participants who consent to behavioral data collection online

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Haire, PhD, Principal Investigator — Kirby Institute
Locations (4):
- Australia (4):
  - Royal Prince Alfred Hospital Sexual Health Medicine, Camperdown, New South Wales
  - Sydney Sexual Health Centre, Sydney, New South Wales
  - Kirketon Road Centre, Sydney, New South Wales
  - Melbourne Sexual Health Centre, Melbourne, Victoria